CLINICAL TRIAL: NCT02213549
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Determine the Effect of Ume Paste and Ginger Powder in Prediabetic Subjects.
Brief Title: Effect of Coadministration of Ume Paste (Prunus Mume) and Ginger Powder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: KAWAMOTO FOODS CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-996
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 3 placebo capsules/day for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Ume paste and ginger powder (Experimental): 3 experimental capsules/day for 12 weeks.
  Interventions: Dietary Supplement: Ume paste and ginger powder

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Ume paste and ginger powder
  Arms: Ume paste and ginger powder

SUMMARY:
This study is designed to evaluate the effect of ume paste and ginger powder on glucose metabolism in prediabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose 105-125 mg/dL

Exclusion Criteria:

* Taking anti-diabetic drugs
* Taking drugs or functional food that may affect blood glucose level
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease
* History of severe disease and/or major surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose from baseline | Every 6 weeks (Overall 12 weeks)
Change in 2h glucose concentration after the oral glucose tolerance test (OGTT) from baseline | Weeks 0 and 12

SECONDARY OUTCOMES:
Change in HbA1c from baseline | Weeks 0 and 12
Change in glycoalbumin from baseline | Weeks 0 and 12
Change in fasting insulin from baseline | Weeks 0 and 12
Change in homeostasis model assessment-insulin resistance (HOMA-R) from baseline | Weeks 0 and 12
  HOMA-R is calculated as fasting insulin (mU/mL) x fasting glucose (mg/dL) / 405
Change in serum total cholesterol from baseline | Every 6 weeks (Overall 12 weeks)
Change in serum LDL cholesterol from baseline | Every 6 weeks (Overall 12 weeks)
Change in serum HDL cholesterol from baseline | Every 6 weeks (Overall 12 weeks)
Change in serum triglyceride from baseline | Every 6 weeks (Overall 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan